CLINICAL TRIAL: NCT05351476
Title: Resistance Training Modulation of Fat Metabolism in Obese Postmenopausal Women
Brief Title: Exercise Training and Fat Metabolism in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Pennington Biomedical Research Center (Other); University of Arkansas (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00001939; R01DK125728 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Postmenopausal Symptoms; Obesity; Prediabetic State
Keywords: Resistance Exercise; Fat Metabolism; Postmenopause
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Exercise (Experimental): Participants do regular resistance exercise for 12 weeks.
  Interventions: Behavioral: Resistance Exercise
- Endurance Exercise (Experimental): Participants do regular endurance exercise for 12 weeks.
  Interventions: Behavioral: Endurance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — 300 Kcal worth of weight lifting, 3 times/week for 12 weeks
  Other Names: Weight Lifting
  Arms: Resistance Exercise
Behavioral: Endurance Exercise — 300 Kcal worth of treadmill walking, 3 times/week for 12 weeks
  Other Names: Aerobic Exercise
  Arms: Endurance Exercise

SUMMARY:
Adipose tissue turnover plays a critical role in body weight maintenance, and obesity is underscored by the dysregulated balance between fat breakdown and synthesis. Although there are clear health-related benefits of physical activity, little is known about how resistance exercise, as opposed to endurance exercise, can reduce the risk of metabolic disorders, particularly in women. The goal of the proposed study is to investigate the effectiveness of resistance training to improve basal and stimulated fat metabolism in postmenopausal women with obesity and pre-diabetes, potentially serving as a viable and practical approach to prevent the onset of type 2 diabetes.

DETAILED DESCRIPTION:
The primary objective is to compare the effects of 12 weeks of resistance training to endurance training with respect to whole-body and regional lipolytic (fat breakdown) responses to acute walking exercise, (Aim 1), local adrenergic receptor blockade (Aim 2) and in response to insulin during a hyperinsulinemic-euglycemic clamp (Aim 3). The investigators will study the lipolytic response in the context of acute exercise, whole-body fat oxidation and resting energy expenditure data. The investigators will collect data on chronic lipogenesis (fat synthesis) and adipogenesis (fat cell formation), as well as on ambulatory blood glucose control. Microdialysis techniques will be utilized to determine the lipolytic rate in subcutaneous abdominal and gluteal adipose tissue at rest, as well as during and after physical activity (walking) or during a hyperinsulinemiceuglycemic clamp (including thigh muscle), before and after 12 weeks of either resistance training or endurance training. To investigate the adrenergic regulation of lipolysis before, during, and after exercise, a saline/ ethanol solution will be perfused (to monitor blood flow) through three separate microdialysis probes in subcutaneous abdominal and gluteal adipose tissue. The perfusate in the probes will consist of either: 1) no additional substances (control probe) to address Aim 1; or 2) phentolamine, an alpha adrenoreceptor blocker (treatment probe), and 3) propranolol, a beta adrenoreceptor blocker (second treatment probe) to address Aim 2. Hyperinsulinemic-euglycemic clamps will be performed to study the whole-body (with stable isotope tracers) and regional (with microdialysis) antilipolytic effect of insulin, as well as to measure insulin sensitivity with respect to glucose metabolism, before and after the training programs for Aim 3. Immediately following the controlled laboratory experiments, glycerol profiles (index of lipolysis) and glucose profiles (index of glucose control) will continue to be monitored in the participant's free-living environment over the ensuing 18 hours until the following morning. Additionally, at weeks 4 and 12 participants will come to the lab for adipose tissue biopsies of the abdominal and gluteal adipose tissue for determination of adipogenesis and lipogenesis using stable-isotope-labeled water they will drink daily over this eight-week labeling period. Additional measures of fat oxidation as well as chronic and acute fat deposition will allow interpretation of lipolysis in the context of fat oxidation and fat accumulation, while 24-hour lipolysis and glucose profile measures will allow investigation of fat metabolism and glucose control in a free-living condition. These studies will provide a greater understanding of how these exercise modalities affect metabolism in women with obesity and prediabetes, allowing practitioners to make more evidence based exercise prescriptions intended to improve body composition, glycemic control, and weight management.

The sample size for these studies will consist of 120 participants that will be randomly assigned via computer randomization to either resistance training (n=60) or endurance training (n=60) for 12 weeks. This sample size gives sufficient statistical power to detect differences in lipolytic rate and other outcome variables, as determined by previous studies examining similar outcome measures. A combination of stable tracers will be infused into the bloodstream to examine various measures of fat metabolism under resting and exercise conditions, as well as during a procedure that mimics a meal (hyperinsulinemic-euglycemic clamp). However, these various tracers can interfere with each other if studied altogether. Therefore these respective isotope tracer measures will be run in only one-half of the participants from each Aim. 30 participants in the endurance training group and 30 participants in the resistance training group will complete Aims 1 and 2. A different 30 participants in the endurance training group and 30 in the resistance training group will complete Aim 3. Among the 60 participants (30 from each exercise training group) completing Aims 1 and 2, there will be 15 individuals from each exercise training group who will be randomized to undergo the tracer measures during exercise while the other 15 from each exercise training group addressing Aims 1 and 2 will complete the exercise protocol without the tracer methods. These randomization methods will also be applied to the 60 participants completing Aim 3, although these participants will undergo a hyperinsulinemic-euglycemic clamp with or without the tracer methods.

Participants will be recruited, screened, enrolled, and tested during months 4-55 of this grant. Participant recruitment procedures and procurement of needed supplies will occur during the first 3 months of the project. Additional recruitment, as well as screening and testing of participants will occur at 1-2 per month over the ensuing 52 months. Two microdialysis experiments will be performed on participants, one before and one after 12 weeks of exercise training, for a total of 240 microdialysis experiments. This plan will therefore require 4-5 microdialysis tests per month on average during the testing months. Stable label palmitate and glycerol isotope experiments will be conducted in 30 of the 60 participants undergoing the acute walking microdialysis experiments and in 30 of the 60 participants undergoing the clamp experiment. Deuterium water isotope experiments (studies of lipogenesis and adipogenesis) will be conducted in 60 of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Postmenopausal (50-75 yrs.)
* Obese (BMI 30-50 kg/m2)
* Prediabetes (HbA1c 5.7 - 6.4% or fasting blood glucose 100 to 125 mg/dL, or 2hr OGTT blood glucose 140 to 199 mg/dL)
* Sedentary (not performing purposeful exercise training more than 20 minutes per day twice a week)
* Non-smokers
* No hormone replacement therapy for at least the past two years.

Exclusion Criteria:

* Engaging in purposeful resistance training or endurance training (> 20min/day, > 2 days/week)
* Resting blood pressure above 140 mmHg systolic or 90 mmHg diastolic
* Type 1 or type 2 diabetes
* Medical problems in which exercise is contraindicated, such as chronic infections
* History of, or currently presentation with, cancer, cardiovascular or respiratory disease
* Uncontrolled thyroid dysfunction, liver or renal dysfunction
* Taking any medication affecting lipid metabolism
* Musculoskeletal disease or injury that would otherwise prevent engagement in resistance and endurance training
* Smokers and those with diagnosed eating disorders

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline subcutaneous abdominal adipose tissue glycerol concentration at 12 weeks | 12 weeks of resistance or endurance training
  Changes in physical activity (walking)-stimulated lipolysis will be assessed as measured by glycerol concentration in dialysate samples from subcutaneous abdominal adipose tissue utilizing a powerful in-vivo microdialysis methodology
Change from baseline gluteal adipose tissue glycerol concentration at 12 weeks | 12 weeks of resistance or endurance training
  Changes in physical activity (walking)-stimulated lipolysis will be assessed as measured by glycerol concentration in dialysate samples from gluteal adipose tissue utilizing a powerful in-vivo microdialysis methodology
Change from baseline whole-body lipolysis at 12 weeks | 12 weeks of resistance or endurance training
  Whole body lipolysis will be measured using whole body rate of appearance of 2H5-glycerol in blood samples collected at rest, during walking exercise, and for 120 minutes after exercise.

SECONDARY OUTCOMES:
Change in blood flow as measured by ethanol concentrations in dialysate samples from subcutaneous abdominal adipose tissue | 12 weeks of resistance or endurance training
  Ethanol (~10 mM) will be included with the perfusion medium through the microdialysis probe. Blood flow will be expressed as a ratio of the ethanol concentration in the dialysate (outflow) and the ethanol concentration in the perfusate (inflow)
Change in dialysate ethanol data in subcutaneous gluteal adipose tissue | 12 weeks of resistance or endurance training
  Ethanol (~10 mM) will be included with the perfusion medium through the microdialysis probe. Blood flow will be expressed as a ratio of the ethanol concentration in the dialysate (outflow) and the ethanol concentration in the perfusate (inflow)
Change in the ratio of 13CO2 to 12CO2 in breath samples | 12 weeks of resistance or endurance training
  This measure will allow for the calculation of whole-body fat oxidation under conditions of rest, walking exercise, and hyperinsulinemiceuglycemic clamp.
change in body composition | 12 weeks of resistance or endurance training
  Body composition (body mass, lean mass, fat mass, visceral fat) will be measured before and after 12 weeks of resistance or endurance training.
Change in blood growth hormone concentrations | 12 weeks of resistance or endurance training
  Concentrations of growth hormone in plasma samples will be measured before and after 12 weeks of resistance or endurance training.
Change in lipogenesis | 12 weeks of resistance or endurance training
  Fat synthesis will be assessed in fat biopsies from subcutaneous abdominal and gluteal adipose tissue using deuterium labeled fatty acids following deuterated water administration in the free-living setting.
Change in adipogenesis | 12 weeks of resistance or endurance training
  New fat cell formation/proliferation will be assessed in fat biopsies from subcutaneous abdominal and gluteal adipose tissue via adipocytes and preadipocytes DNA quantification using deuterated water in the free-living setting.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Hickner, PhD, Principal Investigator — Florida State University; Michael J Ormsbee, PhD, Principal Investigator — Florida State University; Mostafa M Ali, PhD, Study Director — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonafiglia JT, Rotundo MP, Whittall JP, Scribbans TD, Graham RB, Gurd BJ. Inter-Individual Variability in the Adaptive Responses to Endurance and Sprint Interval Training: A Randomized Crossover Study. PLoS One. 2016 Dec 9;11(12):e0167790. doi: 10.1371/journal.pone.0167790. eCollection 2016. PMID 27936084
- [Background] Kim J, Wang Z, Heymsfield SB, Baumgartner RN, Gallagher D. Total-body skeletal muscle mass: estimation by a new dual-energy X-ray absorptiometry method. Am J Clin Nutr. 2002 Aug;76(2):378-83. doi: 10.1093/ajcn/76.2.378. PMID 12145010
- [Background] Hopkins WG. Measures of reliability in sports medicine and science. Sports Med. 2000 Jul;30(1):1-15. doi: 10.2165/00007256-200030010-00001. PMID 10907753
- [Background] Culver AL, Ockene IS, Balasubramanian R, Olendzki BC, Sepavich DM, Wactawski-Wende J, Manson JE, Qiao Y, Liu S, Merriam PA, Rahilly-Tierny C, Thomas F, Berger JS, Ockene JK, Curb JD, Ma Y. Statin use and risk of diabetes mellitus in postmenopausal women in the Women's Health Initiative. Arch Intern Med. 2012 Jan 23;172(2):144-52. doi: 10.1001/archinternmed.2011.625. Epub 2012 Jan 9. PMID 22231607
- [Background] Kim JY, Hickner RC, Cortright RL, Dohm GL, Houmard JA. Lipid oxidation is reduced in obese human skeletal muscle. Am J Physiol Endocrinol Metab. 2000 Nov;279(5):E1039-44. doi: 10.1152/ajpendo.2000.279.5.E1039. PMID 11052958
- [Background] Hickner RC, Racette SB, Binder EF, Fisher JS, Kohrt WM. Suppression of whole body and regional lipolysis by insulin: effects of obesity and exercise. J Clin Endocrinol Metab. 1999 Nov;84(11):3886-95. doi: 10.1210/jcem.84.11.6137. PMID 10566624
- [Background] Hickner RC, Racette SB, Binder EF, Fisher JS, Kohrt WM. Effects of 10 days of endurance exercise training on the suppression of whole body and regional lipolysis by insulin. J Clin Endocrinol Metab. 2000 Apr;85(4):1498-504. doi: 10.1210/jcem.85.4.6550. PMID 10770188
- [Background] Sial S, Coggan AR, Hickner RC, Klein S. Training-induced alterations in fat and carbohydrate metabolism during exercise in elderly subjects. Am J Physiol. 1998 May;274(5):E785-90. doi: 10.1152/ajpendo.1998.274.5.E785. PMID 9612234
- [Background] Hickner RC, Rosdahl H, Borg I, Ungerstedt U, Jorfeldt L, Henriksson J. The ethanol technique of monitoring local blood flow changes in rat skeletal muscle: implications for microdialysis. Acta Physiol Scand. 1992 Sep;146(1):87-97. doi: 10.1111/j.1748-1716.1992.tb09396.x. PMID 1442130
- [Background] Pierce JR, Maples JM, Hickner RC. IL-15 concentrations in skeletal muscle and subcutaneous adipose tissue in lean and obese humans: local effects of IL-15 on adipose tissue lipolysis. Am J Physiol Endocrinol Metab. 2015 Jun 15;308(12):E1131-9. doi: 10.1152/ajpendo.00575.2014. Epub 2015 Apr 28. PMID 25921578
- [Background] Gavin KM, Cooper EE, Raymer DK, Hickner RC. Estradiol effects on subcutaneous adipose tissue lipolysis in premenopausal women are adipose tissue depot specific and treatment dependent. Am J Physiol Endocrinol Metab. 2013 Jun 1;304(11):E1167-74. doi: 10.1152/ajpendo.00023.2013. Epub 2013 Mar 26. PMID 23531620
- [Background] Ormsbee MJ, Choi MD, Medlin JK, Geyer GH, Trantham LH, Dubis GS, Hickner RC. Regulation of fat metabolism during resistance exercise in sedentary lean and obese men. J Appl Physiol (1985). 2009 May;106(5):1529-37. doi: 10.1152/japplphysiol.91485.2008. Epub 2009 Mar 5. PMID 19265063
- [Background] Ormsbee MJ, Clapper JA, Clapper JL, Vukovich MD. The impact of varying dietary protein on serum IGF-I, IGFBP-1, and IGFBP-3 during 6 days of physical activity. Int J Sport Nutr Exerc Metab. 2007 Apr;17(2):127-39. doi: 10.1123/ijsnem.17.2.127. PMID 17507738